CLINICAL TRIAL: NCT06862453
Title: Safety, Tolerability and Efficacy Against Controlled Human Malaria Infection of PfSPZ-LARC2 Vaccine in Malaria-naïve Adults
Acronym: LARC-Tu
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: Universitätsklinikum Tübingen, Institut für Tropenmedizin Wilhelmstrasse (Unknown); UCLA David Geffen School of Medicine and Fielding School of Public Health (Unknown); Stanford University (Other); Leiden University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DESPZL1
Record Dates: First submitted 2025-03-02; First posted 2025-03-06 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Malaria Falciparum
Keywords: malaria; Plasmodium falciparum; PfSPZ-LARC2 Vaccine
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: This is a first-in-humans, randomized, double-blind, placebo-controlled, single-center Phase 1 clinical trial in two parts, with the performance of Part B conditional on the outcome of Part A.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Access to the unblinded randomization list will be limited exclusively to the syringe preparation team (Pharmaceutical Operations team) and the independent statistician(s) at the data management vendor. These individuals will be unblinded and will not be involved in evaluation or care of the study participants. A copy of participant treatment assignments will be retained at the site in a secure file by the unblinded Pharmaceutical Operations staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A Sentinel Group PfSPZ-LARC2 (Experimental): A sentinel group of 5 volunteers in part A that receives a single dose of 2x10^5 PfSPZ of PfSPZ-LARC2 Vaccine by direct venous inoculation (DVI) on Day 1, will be followed for 28 days (to Day 29) to identify any breakthrough infections.
  Interventions: Biological: PfSPZ-LARC2 Vaccine
- Part A Main Cohort PfSPZ-LARC2 verum group (Experimental): If there are no breakthrough infections by Day 29 in the sentinel, the verum group in the main cohort (n = 18) will undergo immunization. Participants will receive 2x10^5 PfSPZ of PfSPZ-LARC2 Vaccine per immunization dose by DVI. All of the participants in the main cohort will progress through a 3-dose immunization regimen with 2x10^5 PfSPZ of PfSPZ-LARC2 Vaccine administered on Days 1, 6 and 29. Twelve weeks after the third immunization dose, the main cohort participants will undergo homologous CHMI using DVI of 3.2x10^3 PfSPZ of PfSPZ Challenge (NF54).
  Interventions: Biological: PfSPZ-LARC2 Vaccine; Biological: PfSPZ Challenge (NF54)
- Part A Main Cohort Normal Saline control group (Placebo Comparator): The blinded control group (n = 6) of the main cohort will receive normal saline as placebo, also by DVI. All of the participants in the main cohort will progress through a 3-dose immunization regimen of normal saline administered on Days 1, 6 and 29. Twelve weeks after the third immunization dose, the main cohort participants will undergo homologous CHMI using DVI of 3.2x10^3 PfSPZ of PfSPZ Challenge (NF54).
  Edit
  Interventions: Other: Normal Saline (Placebo); Biological: PfSPZ Challenge (NF54)
- Part B Sentinel Group PfSPZ-LARC2 (Experimental): If any vaccinee in Part A develops Pf parasitemia following CHMI, and if the safety monitoring committee (SMC) has recommended that the study should continue, the study will proceed to Part B in which the dose of PfSPZ-LARC2 Vaccine will be doubled to 4x10^5 PfSPZ. A sentinel group of 5 volunteers in part B that receives a single dose of 4x10^5 PfSPZ of PfSPZ-LARC2 Vaccine by direct venous inoculation (DVI) on Day 1, will be followed for 28 days (to Day 29) to identify any breakthrough infections.
  Interventions: Biological: PfSPZ-LARC2 Vaccine
- Part B Main Cohort PfSPZ-LARC2 verum group (Experimental): If there are no breakthrough infections by Day 29 in the sentinel, the verum group in the main cohort (n = 18) will undergo immunization. Participants will receive 4x10^5 PfSPZ of PfSPZ-LARC2 Vaccine per immunization dose by DVI. All of the participants in the main cohort will progress through a 3-dose immunization regimen with 4x10^5 PfSPZ of PfSPZ-LARC2 Vaccine administered on Days 1, 6 and 29. Twelve weeks after the third immunization dose, the main cohort participants will undergo homologous CHMI using DVI of 3.2x10^3 PfSPZ of PfSPZ Challenge (NF54).
  Interventions: Biological: PfSPZ-LARC2 Vaccine; Biological: PfSPZ Challenge (NF54)
- Part B Main Cohort Normal Saline control group (Placebo Comparator): The blinded control group (n = 6) of the main cohort will receive normal saline as placebo, also by DVI. All of the participants in the main cohort will progress through a 3-dose immunization regimen of normal saline administered on Days 1, 6 and 29. Twelve weeks after the third immunization dose, the main cohort participants will undergo homologous CHMI using DVI of 3.2x10^3 PfSPZ of PfSPZ Challenge (NF54).
  Interventions: Other: Normal Saline (Placebo); Biological: PfSPZ Challenge (NF54)

INTERVENTIONS:
Other: Normal Saline (Placebo) — The blinded control group (n = 6) of the main cohort will receive normal saline as placebo, also by DVI.
  Arms: Part A Main Cohort Normal Saline control group; Part B Main Cohort Normal Saline control group
Biological: PfSPZ-LARC2 Vaccine — Plasmodium falciparum (Pf) sporozoite (SPZ) late-arresting replication-competent (LARC) malaria vaccine (PfSPZ-LARC2 Vaccine) contains a deletion of two genes, the Mei2 and LINUP genes, and undergoes developmental arrest in the late liver stages without releasing merozoites into the blood stream (blood stage parasites).
  Arms: Part A Main Cohort PfSPZ-LARC2 verum group; Part A Sentinel Group PfSPZ-LARC2; Part B Main Cohort PfSPZ-LARC2 verum group; Part B Sentinel Group PfSPZ-LARC2
Biological: PfSPZ Challenge (NF54) — Main cohort participants will undergo homologous CHMI using DVI of 3.2x10^3 PfSPZ of PfSPZ Challenge (NF54), which are infectious cryopreserved Pf sporozoites.
  Arms: Part A Main Cohort Normal Saline control group; Part A Main Cohort PfSPZ-LARC2 verum group; Part B Main Cohort Normal Saline control group; Part B Main Cohort PfSPZ-LARC2 verum group

SUMMARY:
This is a first-in-human, randomized, double-blind, placebo-controlled Phase 1 trial of Plasmodium falciparum (Pf) sporozoite (SPZ) late-arresting replication-competent (LARC) malaria vaccine (PfSPZ-LARC2 Vaccine) administered to healthy, malaria-naive study participants in Germany by direct venous inoculation (DVI) to determine safety, tolerability, and vaccine efficacy (VE) against controlled human malaria infection (CHMI). PfSPZ-LARC2 Vaccine contains a deletion of two genes, the Mei2 and LINUP genes, and undergoes developmental arrest in the late liver stages without releasing merozoites into the blood stream (blood stage parasites).

The primary objective of the study is to assess the safety and tolerability of administration of PfSPZ-LARC2 Vaccine, with special attention to the adequacy of attenuation, in the intention-to-treat (ITT) population.

Studies of PfSPZ-LARC2 in FRG mice indicate that Plasmodium falciparum LARC2 parasites halt development in their late liver life cycle stages and do not generate viable merozoites able to initiate blood stage infection. Attenuation in this assay system has been a good predictor of attenuation in humans, indicating that blood stage infection in this trial of PfSPZ-LARC2 Vaccine will not occur. Recent data from Leiden University where a Mei2 single deletion parasite was administered to human participants by mosquito bite confirmed that removing this single gene by itself confers complete attenuation. PfSPZ-LARC2 Vaccine has both Mei2 and LINUP deleted, so it should be completely attenuated.

In order to better understand what side effects might look like, on the small chance that PfSPZ-LARC2 Vaccine is not adequately attenuated, it is important to briefly describe the safety data from studies of PfSPZ-CVac (chloroquine), a whole Plasmodium falciparum sporozoite (PfSPZ) immunization approach that uses cGMP produced, aseptic, purified, cryopreserved, non-attenuated, fully infectious PfSPZ administered under chloroquine cover. This is because the safety and tolerability data from PfSPZ-CVac represent a worst case scenario for what could happen with PfSPZ-LARC2 Vaccine with respect to safety and tolerability, as recipients of PfSPZ-CVac always have blood stage infection after the first immunization, even if small doses are administered. The current standard regimen in malaria-naive adults receiving PfSPZ-CVac is 2.0x10^5 PfSPZ, 62.5-fold higher than the 100% infective dose for controlled human malaria infection (CHMI) in malaria-naive individuals, which is 3.2x10^3 PfSPZ. The blood stage infection is detectable by ultrasensitive qPCR on days 7 to 9 after PfSPZ administration and then clears due to the schizonticidal action of chloroquine. Doses used for PfSPZ-CVac have been escalated to as high as 2x10^5 PfSPZ in malaria-naive adults and 4.0x10^5 PfSPZ in malaria-exposed adults, and are generally well tolerated; however, some individuals experienced symptoms of malaria on days 7 and 8 during the period of transient parasitemia, including Grade 3 adverse events, which can largely be prevented by the administration of drugs such as ibuprofen, naproxen or acetaminophen starting the morning of day 7 or after symptoms appear. Once the first dose of 2x10^5 PfSPZ is administered, immunity develops rapidly, and when the second and third doses are administered at 4-week intervals, there have been no Grade 3 adverse events recorded even in the absence of ibuprofen, naproxen or acetaminophen.

These data from PfSPZ-CVac are relevant because they represent a possible worst-case scenario for PfSPZ-LARC2 Vaccine. In other words, even if the attenuation of PfSPZ-LARC2 parasites is not realized in vivo, the density of parasitemia should not be any higher nor the tolerability any worse than what has already been experienced with non-attenuated PfSPZ-CVac administered at the same PfSPZ dose. On the contrary, we would expect the percentage of participants with a blood stage infection to be lower following PfSPZ-LARC2 Vaccine administration due to its intrinsic attenuation than with non-attenuated PfSPZ, and in individuals with a blood stage infection, the numbers of parasites released from the liver to be lower than with non-attenuated PfSPZ.

This will be the first assessment of PfSPZ-LARC2 Vaccine in humans. While we anticipate that vaccine efficacy (VE) in humans will be similar to that of PfSPZ-CVac, we have no data at this point, and it will be important to collect these comparative data. However, in the Leiden trial, where the Mei2 single knockout called GA2 was administered by mosquito bite, there was good protection after 3 immunizations by exposure to 50 infected mosquitoes (8/9 participants protected against homologous CHMI using 5 infected mosquitoes).

DETAILED DESCRIPTION:
This is a first-in-humans, randomized, double-blind, placebo-controlled, single-center Phase 1 clinical trial in two parts, with the performance of Part B conditional on the outcome of Part A.

In Part A, eligible healthy participants (N = 5) will be enrolled as a sentinel group that receives a single dose of 2x105 PfSPZ of PfSPZ-LARC2 Vaccine by direct venous inoculation (DVI) on Day 1 and will be followed for 28 days (to Day 29) to identify any breakthrough infections. If there are no breakthrough infections by Day 29, the main cohort (n = 24) will undergo immunization. Participants in the verum group (n = 18) of the main cohort will also receive 2x10^5 PfSPZ of PfSPZ-LARC2 Vaccine per immunization dose by DVI. The blinded control group (n = 6) of the main cohort will receive normal saline as placebo, also by DVI. All of the participants in the main cohort will progress through a 3-dose immunization regimen with 2x10^5 PfSPZ of PfSPZ-LARC2 Vaccine or normal saline administered on Days 1, 6 and 29.

Participants in both the sentinel group and main cohort will be followed up for parasitemia and adverse events after immunization. After the first immunization on Day 1 in the sentinel group, qPCR will be performed to monitor for P. falciparum blood stage infections daily from Day 7 (day +6) to Day 21 (day +20) and then every other day to Day 29 (day +28) when terminal treatment begins. Thick blood smears (TBS) to monitor for blood stage parasitemia by microscopy will be made on the days that qPCR is performed and read in real-time. TBS will also be done whenever the physician investigator requests a rapid diagnostic test (for whatever reason).

If blood stage parasitemia is not detected during 28 days of follow-up of the sentinel group, the participants will be treated presumptively under direct observation with a three day regimen of atovaquone-proguanil or artemether-lumefantrine), to assure malaria-free status at the end of their participation in the trial.

As soon as the Day 29 qPCR of the sentinel volunteers is determined to be negative, the 24 participants of the main cohort may receive their first immunization with PfSPZ-LARC2 Vaccine or placebo. Following a first immunization on Day 1, the main cohort will receive a second immunization five days later, on Day 6. The qPCR follow-up for the first immunization begins on the next day (Day 7) and will be performed daily from Day 7 (day +6) to Day 12 (day +11), then every other day to Day 22 (day +21) and then weeky thereafter until four weeks after the third immunization, noting that the chance of breakthrough should be much reduced after the first and second immunizations due to the development of immunity. TBS will be performed concurrently as described above and read in real-time.

Twelve weeks after the third immunization dose, the 24 main cohort participants will undergo homologous CHMI using DVI of 3.2x103 PfSPZ of PfSPZ Challenge (NF54). The follow-up for CHMI is described below.

The outcome of CHMI will determine what is done for Part B. As the goal is to achieve 100% protection against homologous CHMI at 12 weeks (this parallels what 2x10^5PfSPZ of PfSPZ-CVac (chloroquine) achieved against heterologous CHMI using the same dose of PfSPZ), if any vaccinee in Part A develops Pf parasitemia following CHMI, and if the safety monitoring committee (SMC) has recommended that the study should continue, the study will proceed to Part B in which the dose of PfSPZ-LARC2 Vaccine will be doubled to 4x10^5 PfSPZ. In other respects, Part B will be the same as Part A, with a sentinel group receiving one dose, and the main cohort three doses on Days 1, 6 and 29, and all 24 participants from the main cohort undergoing CHMI 12 weeks later using standard DVI of 3.2x10^3 PfSPZ of PfSPZ Challenge (NF54) as in Part A.

The rationale for Part B is that protection may be improved by using a higher dose for immunization. This dose of 4x10^5 PfSPZ has been administered using the fully infectious, non-attenuated PfSPZ of PfSPZ-CVac to 158 adult Africans and was well tolerated. Moreover, doses of fully attenuated (irradiated) PfSPZ as high as 2.7x10^6 - 6.75-fold higher than the 4x10^5 PfSPZ dose proposed here - have been administered to both malaria-naive and malaria-exposed adults and were well tolerated. Thus, we do not expect safety issues to be associated with this dose.

Definition of blood stage parasitemia during the immunization phase: qPCR following immunization may be transiently positive early on during follow-up by detecting circulating parasite nucleic acids released from infected hepatocytes, even if there are no viable parasites released into the blood. Thus, an early positive qPCR signal will not be considered an indication of presence of blood stage parasite infection. Rather, the trial will require a qPCR signal that crosses a pre-determined threshold of 1x10^2 parasites/mL on one qPCR result and then registers an at-minimum 4 times higher value on a subsequent result after at least 48 hours to be recognized as failure in genetic attenuation of PfSPZ-LARC2 Vaccine. This will be counted as blood stage infection whether or not the participant experiences symptoms. A positive TBS will also be considered an indication of blood stage parasite infection.

In case of blood stage infection during immunization phase: If the qPCR threshold for blood stage infection is met in any participants or a TBS is positive, they will be treated. The SMC and the clinical and IND Sponsors will be convened. The SMC, Clinical Sponsor and IND Sponsor will decide on the continuation of the study participant with immunization and/or CHMI procedures as well as on the continuation of the overall study.

Additional safety evaluations: Although blood stage infection is the primary focus of the safety evaluation, adverse events will be recorded. Solicited local AEs will be followed for seven days after each immunization, solicited systemic AEs will be followed from the first vaccination until 28 days after the last immunization, and unsolicited AEs will also be followed from the first vaccination until 28 days after the last immunization. In addition, laboratory testing (complete blood count, creatinine, aspartate aminotransferase) will be done before each of the three immunizations and during the follow-up period to assess laboratory abnormalities. Finally, at the day of PfSPZ Challenge administration for CHMI solicited local AEs will be followed for seven days, solicited systemic AEs will be followed for seven days, and unsolicited AEs will be monitored through day +21 to assess the tolerability of any parasitemias that develop in challenged research participants. In addition, during the period of any antimalarial treatment and continuing for three days after the last day of treatment, solicited systemic adverse events will be monitored. Serious adverse events (SAEs) and medically-attended adverse events (MAAEs) will be followed throughout the study.

CHMI and last study visit: The follow-up for CHMI in the main groups will be for 21 days, with daily qPCR and TBS performed from CHMI day +6 to day +21 (corresponds to CHMI Day 7 to CHMI Day 22). Those developing parasitemia by qPCR or TBS will be treated under direct observation with a three day regimen of atovaquone-proguanil or artemether-lumefantrine. Any participant still negative on CHMI day +21 will be treated under direct observation as a safety precaution on CHMI day +21, day +22 and day +23, with the last in-person study visit on day CHMI+23 (corresponds to CHMI Day 24). If qPCR is positive on day +23, however, daily qPCR will continue until there have been two consecutive negative days. There will be one additional study interview six months after last immunization in all groups, which may be done by telephone call, to make sure all participants remain in good health.

Definition of parasitemia during the challenge phase: Parasitemia following CHMI is defined as one qPCR result above 1x10^2 parasites/mL after CHMI with PfSPZ Challenge or a positive TBS.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (male or non-pregnant female) 18 to 45 years of age.
* Able and willing to participate for the duration of the study.
* Able and willing to provide written informed consent.
* Physical examination and laboratory results without clinically significant findings.
* Women of childbearing potential must agree to use effective means of birth control (e.g. oral or implanted contraceptives, IUD, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner) during the entire study.
* Due to the potential for reduced effectiveness of hormonal contraceptives during artemether and/or lumefantrine treatment, participants will be counseled to add an additional barrier method of contraception during treatment.
* Women with a history of surgical or chemical sterilization (e.g. tubal ligation, hysterectomy, other) must provide written documentation of the procedure from a health care provider.
* Agree not to travel to a malaria endemic region during the course of the trial.

Exclusion Criteria:

* Unable to provide informed consent including inability to pass the test of understanding.
* Receipt of a malaria vaccine in a prior clinical trial.
* History of a splenectomy or sickle cell disease.
* History of a neurologic disorder (including non-febrile seizures or complex febrile seizures) or formal history of migraine headache.
* Current use of systemic immunosuppressant pharmacotherapy.
* Receipt of a live vaccine within 4 weeks of first immunization or of 3 or more non-live vaccines within 2 weeks of first immunization.
* Women who are breast-feeding, pregnant or planning to become pregnant during the study period.
* Known allergy or hypersensitivity reaction (e.g., anaphylaxis, erythema multiforme or Stevens-Johnson syndrome, angioedema, vasculitis) to atovaquone-proguanil (Malarone®), artemether-lumefantrine (Coartem®), any components of these formulations, or any component of the investigational products.
* History of anaphylaxis or other life-threatening reaction to a vaccine.
* Participation in any study involving investigational vaccine or drug within 4 weeks prior to enrollment that in the estimation of the site PI might adversely affect the individual's safety or the quality of data to be collected.
* Evidence of increased cardiovascular disease risk; defined as >10% five-year risk by non-laboratory method (Gaziano, 2008) [80].
* Plan to participate in another investigational vaccine/drug research during the study.
* Plan for major surgery between enrollment until 28 days post-CHMI.
* Use or planned use of any drug with anti-malarial activity that would precede or coincide with malaria challenge or vaccination.
* Anticipated use of medications known to cause drug reactions with atovaquone-proguanil or artemether-lumefantrine such as tetracycline, rifampin, rifabutin, cimetidine, metoclopramide, antacids, anti-coagulants such as coumarin, indinavir, and kaolin.
* Anticipated use of medications known to:

  * Be substrates, inhibitors or strong inducers of CYP3A4 (e.g., rifampin, carbamazepine, phenytoin, and/or St. John's wort) [strong inducers of CYP3A4 when taken concomitantly with artemether and/or lumefantrine can result in decreased concentration(s) and loss of antimalarial efficacy].
  * Be metabolized by the cytochrome enzyme CYP2D6 (e.g., primaquine, tafenoquine, flecainide, imipramine, amitriptyline, clomipramine).
  * Have a mixed effect on CYP3A4 (e.g., antiretrovirals).
  * Prolong the QT interval (e.g., quinine, quinidine, halofantrine, mefloquine, procainamide, disopyramideamiodarone, sotalol, pimozide, ziprasidone, tetracycline, doxycline, fluoroquinolone, imidazole, and triazole antifungal agents). Note: in the case of halofantrine, this drug may not be used within a month of artemether/lumefantrine due to its very significant effect on QT interval.
* Positive HIV, HBsAg or HCV serology.
* An abnormal electrocardiogram, defined as one showing pathologic Q waves and significant ST-T wave changes; left ventricular hypertrophy; any non-sinus rhythm including isolated premature ventricular contractions, but excluding isolated premature atrial contractions; right or left bundle branch block; or advanced (secondary or tertiary) A-V heart block; or other clinically significant abnormalities on the electrocardiogram.
* History of symptomatic cardiac arrhythmias, with clinically relevant bradycardia or with severe cardiac disease.
* Family history (grandparents, parents or siblings) of congenital prolongation of the QT interval or sudden death.
* History of disturbances of the electrolyte balance (e.g., hypokalemia or hypomagnesemia).
* History of severe renal impairment (creatinine clearance <30 mL/min) (risk of pancytopenia in patients with severe renal impairment treated with proguanil).
* History of chronic liver disease.
* Any clinically significant deviation from the normal range in biochemistry or hematology tests measured at screening and not resolving.
* Any medical, psychiatric, social, behavioral or occupational condition or situation (including active alcohol or drug abuse) that, in the judgment of the site PI, impairs the participant's ability to give informed consent, increases the risk to the participant of participation in the study, affects the ability of the participant to participate fully in the study, or might negatively impact the quality, consistency, integrity or interpretation of data derived from their participation in the study. This includes persons in emergency situations such as refugees.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of administration of PfSPZ-LARC2 Vaccine, with special attention to the adequacy of attenuation, in the intention-to-treat (ITT) population: infection | 28 days after immunization
  Number of trial participants with blood stage infection during the first 28 days after immunization.
Safety and tolerability of administration of PfSPZ-LARC2 Vaccine, with special attention to the adequacy of attenuation, in the intention-to-treat (ITT) population: related AEs | 7 days after injection of PfSPZ-LARC2 Vaccine
  Incidence of at least possibly related grade 3 solicited adverse events (AE) and grade 3 abnormal laboratory values occurring in the 7 days after injection of PfSPZ-LARC2 Vaccine .
Safety and tolerability of administration of PfSPZ-LARC2 Vaccine, with special attention to the adequacy of attenuation, in the intention-to-treat (ITT) population: related SAEs | Time of first immunization to the end of the study
  Incidence of related serious adverse events (SAEs)

SECONDARY OUTCOMES:
Vaccine Efficacy (VE) (1 minus the risk ratio) against homologous CHMI with PfSPZ Challeng(NF54) conducted 12 weeks after 3rd immunization in the modified ITT (mITT) population | 21 days following CHMI
  Proportion of protected volunteers following CHMI. Protection is defined as the absence of parasitemia in the peripheral blood for +21 days following CHMI with PfSPZ Challenge (NF54) in volunteers who received PfSPZ-LARC2 Vaccine.
Humoral immune responses to PfCSP and their relationship to VE. | The day before immunization until 21 days post CHMI
  Antibody responses as measured by PfCSP ELISA.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tubingen, Wilhelmstraße 27, Tubingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided